CLINICAL TRIAL: NCT01070823
Title: JCV Antibody Program in Patients With Relapsing Multiple Sclerosis Receiving or Considering Treatment With Tysabri®: STRATIFY-1
Brief Title: JC-Virus (JCV) Antibody Program
Acronym: STRATIFY-1
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Collaborators: United BioSource, LLC (Industry); Elan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 101JC401
Record Dates: First submitted 2010-02-17; First posted 2010-02-18 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Multiple Sclerosis
Keywords: Sample Collection; JCV; PML
MeSH Terms: conditions — Multiple Sclerosis | interventions — Natalizumab

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Urine and Plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Relapsing Multiple Sclerosis: Participants receiving or considering treatment with Tysabri® (natalizumab).
  Interventions: Drug: Tysabri® (natalizumab)

INTERVENTIONS:
Drug: Tysabri® (natalizumab) — Prescribed according to the TYSABRI Outreach: United Commitment to Health (TOUCH) Prescribing Program
  Other Names: natalizumab; BG0002

SUMMARY:
The primary objective is to define the prevalence of serum anti-JCV antibody in relapsing multiple sclerosis (MS) participants receiving Tysabri® (natalizumab) or being considered for such treatment. Secondary objectives are to analytically validate the anti-JCV antibody assay in a plasma matrix and to determine changes in anti-JCV antibody status over time.

DETAILED DESCRIPTION:
This study requires serum, plasma and urine collection at enrollment and every 6 months thereafter for up two years.

ELIGIBILITY:
Key Inclusion Criteria:

* Relapsing multiple sclerosis (MS) patients interested in or considering beginning treatment with Tysabri® (natalizumab).

Key Exclusion Criteria:

* Patients participating in any other Tysabri® (natalizumab) clinical trial or study sponsored by Biogen Idec or Elan may not participate in this study.

NOTE: Other protocol-defined inclusion/exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with relapsing Multiple Sclerosis (MS) receiving commercial Tysabri® (natalizumab) and patients being considered for such treatment.
Sampling Method: Probability Sample
Enrollment: 1096 (Actual)
Dates: Start 2010-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of serum anti-JC virus (JCV) antibody | Day 1
  Prevalence of anti-JCV antibodies will be estimated as the number of participants with anti-JCV antibodies detected in serum divided by the total number of participants with a serum sample that was evaluated.
Number of participants with a false negative test | Day 1
  Confirm the false negative rate for serum anti-JCV antibody [assay].

SECONDARY OUTCOMES:
Changes in JCV antibody status over time | Every 6 months for 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (11):
- United States (11):
  - Research Site, Aurora, Colorado
  - Research Site, Atlanta, Georgia
  - Research Site, Cullman, Georgia
  - Research Site, Barrington, Illinois
  - Research Site, Brighton, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Raleigh, North Carolina
  - Research Site, Portland, Oregon
  - Research Site, Round Rock, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Milwaukee, Wisconsin